CLINICAL TRIAL: NCT00845494
Title: Efficacy of a Behavioral Based Education Intervention to Decrease Medication History Errors Among Professional Nurses.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Waukesha Memorial Hospital (Other)
Responsible Party: Kathy Becker, PhD(c), MS, RN, Waukesha Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 554
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Medication Errors
Keywords: Medication history; medication errors; Reduction of admission medication history errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- medication history education (Other): Four hospital unit nurses asked to participate in the study. Two nursing units will receive the cognitive behavioral intervention.
  Interventions: Behavioral: cognitive behavioral intervention

INTERVENTIONS:
Behavioral: cognitive behavioral intervention — The intervention will consist of an hour of cognitive behavioral education. The first 15 minutes spent discussing cases examples of medication errors. The next 15 minutes will include identifying old rules or assumptions nurses have about medication history obtainment. The next 15 minutes will be utilized reviewing a medication tool to be used, and the last 15 minutes will be discussing techniques to help nurse obtain information from elderly patients.

SUMMARY:
The purpose of the study is to determine if a behavioral knowledge based education intervention will decrease medication transcription errors among professional nurses when admitting elder patients to a hospital. The hypothesis is those professional nurses who receive the behavioral-cognitive eduction medication taking intervention will have fewer medication errors than those professional nurses who do not.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working 20 hours a week or more

Exclusion Criteria:

* Nurses working less than 20 hours a week
* Nurse working as a float or pool nurse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in medication errors on admission medication history form after intervention | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Waukesha Memorial Hospital, Waukesha, Wisconsin, United States